CLINICAL TRIAL: NCT02861365
Title: Quantitative Myocardial Perfusion, Myocardial Scarring and Their Contribution to Late Clinical Decompensation in Adults With Congenital Heart Disease
Brief Title: Myocardial Perfusion and Scarring in Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Laura Olivieri, MD, Children's National Research Institute
Other Study IDs: Pro00003067; contract (Other: NIH)
Record Dates: First submitted 2016-07-12; First posted 2016-08-10 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of the perfusion of the myocardium in adults with specific forms of repaired congenital heart disease using established cardiac MRI techniques and correlating perfusion with clinical outcomes.

DETAILED DESCRIPTION:
This is a study of the perfusion of the myocardium in adults with specific forms of repaired congenital heart disease using established cardiac MRI techniques and correlating perfusion with clinical outcomes. The investigators objectives are to examine myocardial perfusion both during stress and at rest in adults with repaired or palliated congenital heart disease as well as quantify ventricular function, regional myocardial strain and evidence of myocardial fibrosis with quantitative measures of myocardial perfusion. The specific aim of this study is to understand whether clinical subendocardial perfusion defects contribute to the late decompensation of adult subjects that have single ventricle physiology and adult subjects that have a systemic right ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* All defects that have a right ventricle that supports the systemic circulation
* All defects with a functional single ventricle
* Written informed consent

Exclusion Criteria:

* Subjects with a contraindication to magnetic resonance imaging (MRI) scanning will be excluded. These contraindications include subjects with the following devices:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker or defibrillator
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump
  * Metal shrapnel or bullet
* Severe heart damage that makes it difficult to breathe while lying flat
* Pregnant women (Women of childbearing potential who are uncertain as to whether they are pregnant will be required to have a screening urine or blood pregnancy test)
* Subjects with active symptoms of myocardial ischemia occurring despite maximally tolerated doses of oral antianginal therapy and intravenous nitroglycerin
* Furthermore, the following subject groups will be excluded from studies involving the administration of MRI contrast agents:

  * lactating women unless they are willing to discard breast milk for 24 hours after receiving gadolinium
  * renal disease (estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73 m2 body surface area)

The eGFR will be used to estimate renal function if reported by the laboratory. Otherwise, estimated glomerular filtration rate (eGFR) can be based on the Modification of Diet in Renal Disease (MDRD) study equation (see below) in subjects with stable renal function. This formula is not applicable to subjects with acute renal insufficiency:

eGFR (ml/min/1.73 m2) = 175 x (serum creatinine)-1.154 x (age)-0.203 x 0.742 (if the subject is female) x 1.212 (if the subject is black)

Additional Exclusion Criteria for Vasodilator Stress MRI:

* Myocardial infarction within 24 hours
* Uncontrolled heart failure
* Uncontrolled asthma or emphysema
* Ventricular arrhythmia (sustained ventricular arrhythmia at the time of MR scan)
* Second degree heart block or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Myocardial Ischemia measuring coronary perfusion reserve. | 5 years
  Compare quantitative myocardial perfusion at stress and rest with measures of systolic and diastolic function in exams performed in close temporal proximity.
Myocardial Ischemia measuring ejection fraction. | 5 years
  Compare the extent of myocardial ischemia through ejection fraction measurement of the systemic ventricle.
Myocardial Ischemia measuring heart inflow Doppler. | 5 years
  Compare heart inflow Doppler of the systemic atrioventricular valve to understand the extent of myocardial ischemia.

SECONDARY OUTCOMES:
Scarring and fibrosis by measuring Late Gadolinium Enhancement results. | 5 years
  Directly compare the extent of myocardial scarring/fibrosis with echo-derived measures of systolic and diastolic function.
Scarring and fibrosis by measuring systolic and diastolic function. | 5 years
  Compare the extent of myocardial scarring/fibrosis with echo-derived measures of systolic and diastolic function.
Comparison of MRI measurements with blood test. | 5 years
  Number of participants with predictable future heart failure symptom will be assessed by comparing all cardiac MRI exam measurements with blood test.
Comparison of MRI measurements with walk test. | 5 years
  Number of participants with predictable future heart failure symptom will be assessed by comparing all cardiac MRI exam measurements with walk test.
Comparison of MRI measurements with NY Heart Association class | 5 years
  Number of participants with predictable future heart failure symptom will be assessed by comparing all cardiac MRI exam measurements with NY Heart Association class.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Olivieri, MD, Principal Investigator — Children's National Health Systems
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of MRI scans will be shared with the primary cardiologist.
Supporting Information: CSR
Time Frame: MRI report becomes available once the scan has been assessed, usually within 24 hours. It will be available indefinitely.
Access Criteria: Primary care takers will have access to this report.

REFERENCES:
- [Background] Verheugt CL, Uiterwaal CS, van der Velde ET, Meijboom FJ, Pieper PG, van Dijk AP, Vliegen HW, Grobbee DE, Mulder BJ. Mortality in adult congenital heart disease. Eur Heart J. 2010 May;31(10):1220-9. doi: 10.1093/eurheartj/ehq032. Epub 2010 Mar 5. PMID 20207625
- [Background] Rutledge JM, Nihill MR, Fraser CD, Smith OE, McMahon CJ, Bezold LI. Outcome of 121 patients with congenitally corrected transposition of the great arteries. Pediatr Cardiol. 2002 Mar-Apr;23(2):137-45. doi: 10.1007/s00246-001-0037-8. Epub 2002 Feb 19. PMID 11889523
- [Background] Meijboom F, Szatmari A, Deckers JW, Utens EM, Roelandt JR, Bos E, Hess J. Long-term follow-up (10 to 17 years) after Mustard repair for transposition of the great arteries. J Thorac Cardiovasc Surg. 1996 Jun;111(6):1158-68. doi: 10.1016/s0022-5223(96)70217-9. PMID 8642816